CLINICAL TRIAL: NCT00436891
Title: The Epidemiology of Group A Streptococcal Infections in Fiji (Fiji GrASP) - Part 4 -The Prevalence of Group A Streptococcal Pyoderma and Scabies in Infants in Fiji
Brief Title: Streptococcal Infections in Fiji - Prevalence of Group A Streptococcal Pyoderma and Scabies in Infants in Fiji
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 06-0081; Fiji GrASP Part 4
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2008-05-02 (Estimated); Status verified 2007-10

CONDITIONS: Streptococcus Group A
Keywords: Group A Streptococcus, scabies, pyoderma, Fiji
MeSH Terms: conditions — Scabies; Pyoderma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Group A streptococcus (GAS) is a bacteria that causes many different sicknesses in children and adults. This study will look at the number of cases of pyoderma (bacterial skin infection) and scabies (skin mites that cause itching) in 550 infants 12 months or younger in Fiji. (GAS can cause pyoderma, and sometimes skin sites infested with scabies can become infected with GAS bacteria.) The study will also look at the makeup of GAS and how certain medications affect GAS. The infants will be involved in the study for approximately 1 week. Their skin will be examined for pyoderma and scabies. A swab sample will be taken from the pyoderma area to test for GAS. The researchers hope to see how often these skin infections occur and how they affect the Fijian population. The information will help the researchers to develop better treatment and possibly a vaccine to prevent infection. Infants with pyoderma that is defined as "greater than mild" will be referred for treatment.

DETAILED DESCRIPTION:
Group A beta-hemolytic streptococcus, a common infective agent in children and adults, causes the widest range of clinical disease of any bacterium. This study is the fourth of five studies in a larger project aimed at evaluating the epidemiology of infections caused by the group A streptococcus (GAS) in Fiji. This larger project is called the Fiji Group A Streptococcal Project (Fiji GrASP). Fiji GrASP is in turn part of a larger program aimed at progression of a novel GAS vaccine - this program is the project entitled "Global GAS Vaccine Based on the M-Protein." The three broad aims of the Fiji GrASP epidemiologic studies are: (1) to establish the burden of disease of GAS infections in Fiji; (2) to describe the molecular epidemiology of GAS isolates in Fiji and; (3) to establish natural immunologic correlates of protection of a J8 vaccine if they exist. This is a cross-sectional study of 550 infants over a 2-month period. Skin will be examined for pyoderma and scabies, and swabs will be taken from pyoderma lesions once. All GAS isolates from skin swabs will undergo genetic sequencing of the N-terminal and C-repeat regions (for the J8 epitope) of the M protein at QIMR. One hundred skin swabs will undergo antimicrobial susceptibility testing against penicillin, erythromycin, clindamycin and chloramphenicol. The primary objectives of the study are to estimate the point prevalence of GAS pyoderma in 550 infants in the Central Division of Fiji and to estimate the point prevalence of scabies in 550 infants in the Central Division of Fiji. The secondary objectives of the study are to genotypically characterize group A streptococci isolated from skin swabs from pyoderma lesions in infants in Fiji and to determine antimicrobial susceptibility to penicillin, clindamycin, erythromycin and chloramphenicol in 100 GAS isolates from skin swabs. The primary endpoints of the study are to determine the number of cases of pyoderma and the number of cases of scabies. The secondary endpoints are: (1) to determine the number of children with pyoderma and scabies; (2) to determine the number of GAS isolates from skin swabs that contain the J8 epitope and the overall emm-type distribution of GAS isolates and; (3) to complete antibiograms of GAS isolates from skin to penicillin, clindamycin, erythromycin and chloramphenicol.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent from parents/guardians will be obtained for all study participants.
2. Infants less than or equal to 12 months of age
3. Attending Navua Health Center and/or Raiwaqa/Vatuwaqa Health Centre
4. Infants can only be enrolled on one occasion.

Exclusion Criteria:

1. Subjects greater than 12 months of age

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 550
Dates: Start 2007-02; Study Completion 2007-04

CONTACTS AND LOCATIONS:
Locations (1):
- Colonial War Memorial Hospital, Suva, Fiji